CLINICAL TRIAL: NCT05483296
Title: Modulating Evening Responses to Light by Afternoon Light Exposure in Adolescents
Brief Title: Effects of Afternoon and Evening Light on Teenagers' Melatonin Levels, Alertness, Sleepiness and Sleep
Acronym: TeenLight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Psychiatric Clinics Basel (Network)
Responsible Party: Principal Investigator, Dr Christian Cajochen, Principal Investigator/ Sponsor-Investigator, University Psychiatric Clinics Basel
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2022-00432
Record Dates: First submitted 2022-07-25; First posted 2022-08-02 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy; Teenager; Healthy Lifestyle
Keywords: melatonin; polysomnography; EEG; sleep; afternoon light; pupil size; evening light

STUDY DESIGN:
Intervention Model Description: The protocol is a full within-subject trial (cross-over). All participants will conduct three 18-hour experiment sessions and go through the same protocol except for the sequence of the experiment sessions (counter-balanced and randomised).
Masking Description: Entirely blinding the differences between the experiment's light conditions is unattainable (for both participants and experimenters) because of the visibly perceivable differences in brightness between them. However, the melatonin and objective EEG measurements should not be significantly affected by any expectancy effects. Participants will not be told the expected effects of the different light exposure conditions to minimise the expectancy effects for behavioural measures (i.e., PVT) and subjective measurements. Information on the hypothesized outcomes will be withheld from the volunteers and study helpers until after completing all sessions. During the analysis, light intensity conditions and participant IDs will be coded to withhold information from the analytic team about the light intensity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Crossover sequence 1: Dim, Moderate, Bright (Experimental): All participants will go through all three light conditions in the three experiment sessions: They will receive white fluorescent overhead light (given in melanopic EDI at eye level) as the 4h afternoon light intervention. In the first experimental session, they receive an intensity of <10 lx. In the second experimental session, they receive an intensity of ~100 lx, and in the third experimental session, they receive an intensity of >1000 lx.
  Interventions: Other: Dim light condition; Other: Moderate light condition; Other: Bright light condition
- Crossover sequence 2: Dim, Bright, Moderate (Experimental): All participants will go through all three light conditions in the three experiment sessions: They will receive white fluorescent overhead light (given in melanopic EDI at eye level) as the 4h afternoon light intervention. In the first experimental session, they receive an intensity of <10 lx. In the second experimental session, they receive an intensity of >1000 lx, and in the third experimental session, they receive an intensity of ~100 lx.
  Interventions: Other: Dim light condition; Other: Moderate light condition; Other: Bright light condition
- Crossover sequence 3: Moderate, Dim, Bright (Experimental): All participants will go through all three light conditions in the three experiment sessions: They will receive white fluorescent overhead light (given in melanopic EDI at eye level) as the 4h afternoon light intervention. In the first experimental session, they receive an intensity of ~100 lx. In the second experimental session, they receive an intensity of <10 lx, and in the third experimental session, they receive an intensity of >1000 lx.
- Crossover sequence 4: Moderate, Bright, Dim (Experimental): All participants will go through all three light conditions in the three experiment sessions: They will receive white fluorescent overhead light (given in melanopic EDI at eye level) as the 4h afternoon light intervention. In the first experimental session, they receive an intensity of ~100 lx. In the second experimental session, they receive an intensity of >1000 lx, and in the third experimental session, they receive an intensity of <10 lx.
- Crossover sequence 5: Bright, Moderate, Dim (Experimental): All participants will go through all three light conditions in the three experiment sessions: They will receive white fluorescent overhead light (given in melanopic EDI at eye level) as the 4h afternoon light intervention. In the first experimental session, they receive an intensity of >1000 lx. In the second experimental session, they receive an intensity of ~100 lx, and in the third experimental session, they receive an intensity of <10 lx.
- Crossover sequence 6: Bright, Dim, Moderate (Experimental): All participants will go through all three light conditions in the three experiment sessions: They will receive white fluorescent overhead light (given in melanopic EDI at eye level) as the 4h afternoon light intervention. In the first experimental session, they receive an intensity of >1000 lx. In the second experimental session, they receive an intensity of <10 lx, and in the third experimental session, they receive an intensity of ~100 lx.

INTERVENTIONS:
Other: Dim light condition — During the "Dim" light condition, the four-hour afternoon light exposure at the participants' eye level will be dim (<5 lx melanopic EDI). In the 4.5-hour evening light exposure, this will constitute a light intensity of ~100 lx melanopic EDI at the participants' eye level.
  Arms: Crossover sequence 1: Dim, Moderate, Bright; Crossover sequence 2: Dim, Bright, Moderate
Other: Moderate light condition — During the "Moderate" light condition, the four-hour afternoon light exposure at the participants' eye level will be dim (~100 lx melanopic EDI). In the 4.5-hour evening light exposure, this will constitute a light intensity of ~100 lx melanopic EDI at the participants' eye level.
  Arms: Crossover sequence 1: Dim, Moderate, Bright; Crossover sequence 2: Dim, Bright, Moderate
Other: Bright light condition — During the "Bright" light condition, the four-hour afternoon light exposure at the participants' eye level will be dim (>1000 lx melanopic EDI). In the 4.5-hour evening light exposure, this will constitute a light intensity of ~100 lx melanopic EDI at the participants' eye level.
  Arms: Crossover sequence 1: Dim, Moderate, Bright; Crossover sequence 2: Dim, Bright, Moderate

SUMMARY:
Many teenagers are familiar with this: on school days, they have to get up early; during the day, they hardly get any light exposure; in the evening, they go to bed late - and are then tired at school the next day! Around the world, teenagers are sleep deprived, with studies suggesting that almost half (~45%) suffer from inadequate sleep. Previous investigations have shown that people's sleep-wake rhythm is related to the light conditions that they are exposed to during the day and at night. However, little is known about how different light levels in the afternoon can modulate teenagers' sleep and their bodily responses to light in the late evening. Therefore, the investigators aim to study which lighting conditions have a favourable effect on these aspects and how the potentially harmful effects of light at night can be prevented.

DETAILED DESCRIPTION:
Light exposure during adolescence seems to be the critical component of a vicious circle. Due to the maturation of sleep-wake regulatory systems in combination with progressively ill-timed exposure to light and early school start times, teenagers suffer from the accumulation of sleep depth during school days. Therefore, the proposed study investigates whether the physiological and alerting effects of late evening light exposure in adolescents depend on the intensity of light exposure in the preceding afternoon (primary endpoint: evening melatonin concentration).

The investigators aim to describe dose-response relationships, where the "dose" is the preceding (real-world applicable) afternoon light intensity (< 10 lx, ~100 lx, or >1000 lx EDI, 4-hour duration), and the "responses" are the adolescents' physiological and alerting responses to evening light exposure (~100 lx melanopic EDI, 4.5-hour duration). By this route, the researchers can explore whether increasing afternoon light exposure is a feasible target for ameliorating the detrimental effects of artificial light at night and promoting healthier sleep-wake regulation during adolescence.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Capable of judgment
* Normal BMI (Age-related Body-Mass-Index Percentile > P3 & < P97; approx. corresponding to 28.5 ≥ BMI ≤ 16)
* Signed consent form of participants
* Signed consent form of a legal representative

Exclusion Criteria:

* Pregnancy or breastfeeding (only female)
* Current participation in other clinical trials
* Extreme chronotype (Extreme early or late chronotype/mid sleep time: mid-sleep time < 1:00 / > 7:00)
* Extremely short or long sleep durations during school- or work days (< 6 hours > 11 hours)
* Sleep disorders
* High myopia (< -6 diopters)
* High hyperopia (> +6 diopters)
* Non-normal best-corrected visual acuity (BCVA < 0.5 [20/40])
* General health concerns or disorders, including heart and cardiovascular, neurological, nephrological, endocrinological, and psychiatric conditions
* Ophthalmological or optometric conditions
* Medication impacting visual, neuroendocrine, sleep, and circadian physiology
* Drug and alcohol use (urinary drug screening & breathalyzer test)
* Non-compliance with sleep-wake times: >1 deviation from ±60 minute window sleep and wake-up time
* Non-compliance with caffeine intake (> 1 times caffeine intake)
* Transmeridian travel (>2 time zones) <1 month prior to the first session of the study
* shift work <3 months prior to the beginning of the study

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Salivary melatonin | Through study completion, estimated 1.5 years (within 3 weeks for each participant)
  Salivary melatonin. Saliva samples (>1 mL) will be taken from the participants every 30 Minutes using Salivettes. The Salivettes will be centrifuged, the cotton part removed and immediately frozen at -20°C. At a later point, melatonin [in pg] will be determined in these samples by double-antibody radioimmunoassay (RIA). To quantify melatonin suppression, the analytic team will calculate the area under the curve (AUC) for each laboratory condition.

SECONDARY OUTCOMES:
Sleep Onset Latency (PSG-derived) | Through study completion, estimated 1.5 years (within 3 weeks for each participant)
  The investigators will operationalise Sleep Onset Latency according to the American Academy of Sleep Medicine (AASM) Manual for the Scoring of Sleep and Associated Events (time interval from lights out to the first PSG-derived sleep epoch in minutes).
Slow wave activity (PSG-derived) | Through study completion, estimated 1.5 years (within 3 weeks for each participant)
  The investigators will examine slow-wave activity (SWA; delta power density between 0.5 and 4.5 Hz) during the first sleep cycle. EEG slow-wave activity (SWA) (i.e., delta power density between 0.5 and 4.5 Hz) will be calculated as an indicator of sleep propensity across the night within each non-rapid eye movement NREM part of a sleep cycle.
Sleep stages (PSG-derived) | Through study completion, estimated 1.5 years (within 3 weeks for each participant)
  The investigators will score the PSG-derived sleep stages and arousals according to the American Academy of Sleep Medicine (AASM) Manual for the Scoring of Sleep and Associated Events.
Subjective sleepiness | Through study completion, estimated 1.5 years (within 3 weeks for each participant)
  The investigators will assess subjective sleepiness using the single-item 9-point Karolinska Sleepiness Scale (KSS) - a well-validated, highly sensitive subjective Likert-type measurement scale for subjective sleepiness.
  Scores range from 1 to 9 with higher values on the scale corresponding to higher sleepiness.
Vigilant attention | Through study completion, estimated 1.5 years (within 3 weeks for each participant)
  Objective alertness will be measured using a modified auditory Psychomotor Vigilance Test (aPVT). After a response, the next tone will be played randomly after 2-10 s. The reaction time data will focus on mean 1/reaction time (mean 1/RT), the most sensitive measure for a slight deviation in sleep pressure. Mean 1/RT will be calculated after the removal of false starts and lapses.
Melanopsin sensitivity (pupillary light response) | Through study completion, estimated 1.5 years (within 3 weeks for each participant)
  The investigators will measure changes in the pupil area using silent substitution pupillography and examine the differences between melanopsin response amplitude before the afternoon light condition (pre-light treatment) and the melanopsin response amplitude after the afternoon light condition (post-light treatment).
Skin temperature | Through study completion, estimated 1.5 years (within 3 weeks for each participant)
  Skin temperature will be continuously monitored with six surface temperature thermocouples placed on proximal and distal regions of the body surface. Skin temperatures (distal & proximal) and the distal-proximal skin temperature gradient (DPG) will be calculated.
Objective sleepiness 1 | Through study completion, estimated 1.5 years (within 3 weeks for each participant)
  The volunteers will perform a Karolinska Drowsiness Test (KDT) three times during scheduled wakefulness. During the KDT, participants fixate on a point on the wall from a one-meter distance for five minutes (eyes open). These sessions will provide EEG data with relatively few artefacts. As the first indicator for objective sleepiness, EEG-derived alpha/theta ratio will be calculated.
Objective sleepiness 2 | Through study completion, estimated 1.5 years (within 3 weeks for each participant)
  The volunteers will perform a Karolinska Drowsiness Test (KDT) three times during scheduled wakefulness. During the KDT, participants fixate on a point on the wall from a one-meter distance for five minutes (eyes open). These sessions will provide EEG data with relatively few artefacts. As the second indicator for objective sleepiness, electro-oculogram-derived (EOG-derived) slow-eye movements will be calculated.

OTHER OUTCOMES:
Ambulant light history. | Through study completion, estimated 1.5 years (within 3 weeks for each participant)
  To account for participants' light exposure before they arrive at the experimental site, ambulatory light exposure will be assessed throughout the three weeks of the experiment with actimetry devices (Condor ActTrust). Additionally, participants will be asked to estimate their duration of outdoor light exposure daily. During the experiment, participants will further be instructed to wear a lightweight light sensor.
Actigraphy | Through study completion, estimated 1.5 years (within 3 weeks for each participant)
  Compliance to regular sleep-wake cycles over three weeks will be monitored with the actimetry device starting five days before the first experimental session (baseline + adaptation night) and ending with the final session.
Visual comfort & well-being | Through study completion, estimated 1.5 years (within 3 weeks for each participant)
  An adapted German version of the first six items of the Visual Comfort Scale (VCS) will be used to assess the participant's visual comfort under the different lighting conditions. Additionally, participants will rate their momentary affect and well-being in relation to mood, hunger, relaxation, and motivation. Items are rated on a 7-point Likert-type scale (1-7) with higher values corresponding to a higher manifestation of the characteristic (for instance well-being, the brightness of the light etc.)
Sleep diary | Through study completion, estimated 1.5 years (within 3 weeks for each participant)
  Volunteers will report their sleep and wake episodes using a sleep-wake diary (like a questionnaire).
Sleep quality | Through study completion, estimated 1.5 years (within 3 weeks for each participant)
  In the mornings after the laboratory sleep, participants will additionally fill in a sleep quality questionnaire (Leeds Sleep Evaluation Questionnaire; LSEQ). The LSEQ is a 10-item, subjective, self-report measure that includes a visual analogue scale, where every item is scored from 0 to 10 where 10 corresponds to a higher manifestation of the characteristic (for instance tiredness).
Dream recall | Through study completion, estimated 1.5 years (within 3 weeks for each participant)
  In the mornings after the laboratory sleep, participants will additionally fill in a dream recall questionnaire (Sleep Mentation Questionnaire) which addresses numerous characteristics of dream recall, such as the number of dreams, emotionality, vividness, pleasantness, hostility, and colourfulness, on a Likert-point scale (1: greatly, 2: fairly, 3: little, and 4: not at all). Higher values on the scale correspond to a lower frequency of dreams.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Cajochen, PhD, Principal Investigator — Centre for Chronobiology, University Psychiatric Clinics Basel, Basel, Switzerland
Locations (1):
- Psychiatric University Clinics (UPK), Centre for Chronobiology, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Deidentified, anonymised, non-sensitive data will be made available in a publicly accessible repository hosted on https://figshare.com/ after data collection, curation, and publication. The data will be licensed under Creative Commons Attribution-NonCommercial 4.0 International (CC BY-NC 4.0). This allows for sharing (copying and redistributing the material in any medium or format) and adapting (remixing, transforming, and building upon the material) under the following terms: Users must give appropriate credit, provide a link to the license, and indicate if changes were made. Users may not use the material for commercial purposes. Parts of the anonymised data can become available even before due to journal publications. Therefore, apart from our research team, the dataset might benefit other research groups working on similar questions in the non-visual processing of light.

REFERENCES:
- [Background] Galland BC, Short MA, Terrill P, Rigney G, Haszard JJ, Coussens S, Foster-Owens M, Biggs SN. Establishing normal values for pediatric nighttime sleep measured by actigraphy: a systematic review and meta-analysis. Sleep. 2018 Apr 1;41(4). doi: 10.1093/sleep/zsy017. PMID 29590464
- [Background] Hagenauer MH, Perryman JI, Lee TM, Carskadon MA. Adolescent changes in the homeostatic and circadian regulation of sleep. Dev Neurosci. 2009;31(4):276-84. doi: 10.1159/000216538. Epub 2009 Jun 17. PMID 19546564
- [Background] Lo JC, Lee SM, Lee XK, Sasmita K, Chee NIYN, Tandi J, Cher WS, Gooley JJ, Chee MWL. Sustained benefits of delaying school start time on adolescent sleep and well-being. Sleep. 2018 Jun 1;41(6):zsy052. doi: 10.1093/sleep/zsy052. PMID 29648616
- [Background] Santhi N, Ball DM. Applications in sleep: How light affects sleep. Prog Brain Res. 2020;253:17-24. doi: 10.1016/bs.pbr.2020.05.029. Epub 2020 Jul 25. PMID 32771123
- [Background] Akerstedt T, Gillberg M. Subjective and objective sleepiness in the active individual. Int J Neurosci. 1990 May;52(1-2):29-37. doi: 10.3109/00207459008994241. PMID 2265922
- [Background] Gabel V, Kass M, Joyce DS, Spitschan M, Zeitzer JM. Auditory psychomotor vigilance testing in older and young adults: a revised threshold setting procedure. Sleep Breath. 2019 Sep;23(3):1021-1025. doi: 10.1007/s11325-019-01859-7. Epub 2019 May 8. PMID 31069648
- [Background] Spitschan M, Woelders T. The Method of Silent Substitution for Examining Melanopsin Contributions to Pupil Control. Front Neurol. 2018 Nov 27;9:941. doi: 10.3389/fneur.2018.00941. eCollection 2018. PMID 30538662
- [Background] Parrott AC, Hindmarch I. The Leeds Sleep Evaluation Questionnaire in psychopharmacological investigations - a review. Psychopharmacology (Berl). 1980;71(2):173-9. doi: 10.1007/BF00434408. PMID 6777817
- [Background] Chellappa SL, Munch M, Blatter K, Knoblauch V, Cajochen C. Does the circadian modulation of dream recall modify with age? Sleep. 2009 Sep;32(9):1201-9. doi: 10.1093/sleep/32.9.1201. PMID 19750925